CLINICAL TRIAL: NCT00688818
Title: Randomized, Placebo-Controlled Effectiveness Study of Quetiapine XR in Co-Morbid Depressive and Anxiety Disorders
Brief Title: Quetiapine in Co-Morbid Depressive and Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Arun Ravindran, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 183/2007
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Major Depressive Disorder; Dysthymic Disorder; Anxiety Disorders; Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Post-traumatic Stress Disorder
Keywords: Co-morbid depressive and anxiety disorders; Quetiapine; Randomized; Placebo-controlled; Double-blind; Major depressive disorder; Dysthymic disorder; Anxiety disorders; Generalized anxiety disorder; Social anxiety disorder; Panic disorder; Post-traumatic stress disorder
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Stress Disorders, Post-Traumatic | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine and existing psychotropics (Experimental)
  Interventions: Drug: Quetiapine
- Placebo and existing psychotropics (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine — Patients will be initiated on 50 mg of Quetiapine XR and will be titrated to a maximum dose of 300 mg based on response and tolerability. Dosing will be flexible up to Week 8, and then will remain fixed for until the end of the 12 week period.
  Other Names: Seroquel
  Arms: Quetiapine and existing psychotropics
Drug: Placebo — Patients will be initiated on 50 mg of Placebo and will be titrated to a maximum dose of 300 mg based on response and tolerability. Dosing will be flexible up to Week 8, and then will remain fixed for until the end of the 12 week period.
  Arms: Placebo and existing psychotropics

SUMMARY:
This multi-centred study will be conducted at three centres. The design will be a randomized, placebo-controlled, parallel-group one. This investigation will evaluate the efficacy of add-on Quetiapine XR (extended release) treatment for patients who meet diagnostic criteria for depressive disorders and one or more comorbid anxiety disorder.

DETAILED DESCRIPTION:
The primary objective is to examine the beneficial effect of quetiapine augmentation of first-line antidepressants in refractory depression with co-morbid anxiety, compared to placebo. It is hypothesized that significant improvement on depression and anxiety symptoms will be seen as evidenced by reduction in Hamilton Depression Rating Scale (HAMD-17) and Hamilton Anxiety Scale (HAMA) scores after the 12 week treatment period for those who received Quetiapine XR augmentation compared to those who received placebo.2.2

Secondary objectives: 1) To establish the tolerability and safety of Quetiapine XR versus Placebo in patients with co-morbid depressive and anxiety disorders;2) To assess and compare the efficacy of Quetiapine XR versus Placebo improving quality of life in patients with co-morbid depressive and anxiety disorders.; 3) To assess and compare the efficacy of Quetiapine XR versus Placebo on clinical measures symptoms associated to co-morbid depressive and anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male and female patients must be of 18 to 65 years of age.
* Women of childbearing potential must have a negative pregnancy test and must, in the investigator's opinion, practice a clinically accepted, reliable method of contraception during this study.
* A diagnosis of Major Depressive Disorder or Dysthymic Disorder as defined by DSM-IV criteria and failed to respond to at least one first line treatment. The patient must be receiving antidepressant treatment (SSRIs, SNRIs or mirtazapine).
* A co-morbid diagnosis of one or more of the following: Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, and Post Traumatic Stress Disorder, and Obsessive-Compulsive Disorder, as defined by DSM-IV criteria
* A minimum score of ≥17 at Baseline on the 17-item HAM-D.
* Able to understand and comply with the requirements of the study

Exclusion Criteria:

* The presence or history of Psychotic Disorders, Bipolar Disorders, Mood Disorders with Psychotic Features
* Patients who, in the investigator's judgment, would require treatment with additional psychotherapeutic drugs, electroconvulsive therapy (ECT), or intensive psychotherapy during the course of the study.
* ECT within the preceding 6 months of screening before inclusion.
* Regular, formal psychotherapy (excluding supportive therapy) started within the last 3 months before inclusion.
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate.
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment
* Use of any of the following significant cytochrome P450 inducers in the 14 days preceding enrolment
* Patients who are currently receiving: monoamine oxidase inhibitors, tricyclic antidepressants, oral neuroleptics, or type 1C anti-arrhythmics within two weeks of screening; herbal psychoactive treatments (St. John's Wort, Kava Kava, Gingko Biloba) within two weeks of screening.
* Patients taking SSRIs or SNRIs for less than two weeks or at a less than therapeutic dose prior to enrolment.
* Patients who require concurrent psychotropic medication other than allowed medication specified in protocol.
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation.
* Patients who have met DSM-IV criteria for abuse of or dependence on any drug, including alcohol within 3 months prior to screening.
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
* Patients with clinically significant abnormalities in hematology, clinical chemistry, urinalysis or ECG at the screening visit.
* Involvement in the planning and conduct of the study
* Previous enrolment or randomisation of treatment in the present study.
* Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:a)Unstable DM (HbA1c) >8.5%, b) hospital admission for DM or DM related illness in past 12 weeks, c)not under physician care for DM, d) physician responsible for patient's DM care has not approved patient's participation in the study,or indicated DM is controlled e)change in dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period will not be less than 8 weeks, g)taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks (Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study)
* An absolute neutrophil count (ANC) of <= 1.5 x 10^9 per

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD-17) | 12 weeks

SECONDARY OUTCOMES:
Hamilton Anxiety Scale | Baseline, 6 weeks and 12 weeks
Quality of Life Enjoyment and Satisfaction Scale | Baseline, 6 weeks and 12 weeks
Penn State Worry Questionnaire | Baseline, 6 weeks and 12 weeks
Panic Disorder Severity Scale | Baseline, 6 weeks and 12 weeks
Leibowitz Social Anxiety Scale | Baseline, 6 weeks and 12 weeks
Post-traumatic Diagnostic Scale | Baseline, 6 weeks and 12 weeks
Clinical Global Impression Scale | Baseline, 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arun Ravindran, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (4):
- Canada (4):
  - Chatham-Kent Health Alliance, Chatham, Ontario
  - Centre for Neuropsychiatric Study, Markham, Ontario
  - Credit Valley Medical Arts Centre, Mississauga, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- [Derived] Ravindran N, McKay M, Paric A, Johnson S, Chandrasena R, Abraham G, Ravindran AV. Randomized, Placebo-Controlled Effectiveness Study of Quetiapine XR in Comorbid Depressive and Anxiety Disorders. J Clin Psychiatry. 2022 Mar 21;83(3):21m14096. doi: 10.4088/JCP.21m14096. PMID 35324094
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research